CLINICAL TRIAL: NCT02942810
Title: A Phase 1, Open-label, Single-dose Study to Investigate the Pharmacokinetics of Intravenous WCK 5222 (FEP-ZID) in Patients With Renal Impairment
Brief Title: To Investigate The Pharmacokinetics Of Intravenous WCK 5222 (FEP-ZID) In Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W-5222-102
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — cefepime-zidebactam; Cefepime

ARMS (1):
- WCK 5222 (Cefepime and zidebactam combination) (Experimental): IV infusion over a period of 60 minutes
  Interventions: Drug: WCK 5222

INTERVENTIONS:
Drug: WCK 5222 — IV infusion over a period of 60 minutes
  Other Names: Cefepime and zidebactam combination

SUMMARY:
This is a Phase 1, open label, single-dose, pharmacokinetic study to be conducted in male and female subjects with normal and impaired renal function. The study will be composed of five groups of patients with mild (6 patients), moderate (6 patients), severe (6 patients) renal impairment, end stage renal disease patients on hemodialysis (6 patients) and their respective matched controls in 1:1 ratio (24 healthy subjects with normal renal function). The severity of renal impairment will be assessed based on estimated creatinine clearance (CLCR) by the Cockcroft-Gault equation

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) 18.0 and 40.0 (kg/m2) and body weight of at least 50 kg.

   Patients with renal impairment:
2. Have a diagnosis of renal impairment that has been stable, without any change in overall disease status in the last 1 month

   Healthy Subjects:
3. Have normal renal function with creatinine clearance more than 90 mL/min and no evidence of any disease or condition that may affect pharmacokinetics of FEP ZID.
4. A resting blood pressure 90-145 (systolic) / 60-95 (diastolic) mmHg for healthy volunteers and 90-155 (systolic) / 50-100 (diastolic) mmHg for patients with renal impairment.

Exclusion Criteria:

1. History or presence of significant hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, rheumatologic, hepatic, urologic, immunologic, infectious, skin and subcutaneous tissue, psychiatric or mood disorders (including any past suicide attempt), or uncontrolled metabolic or endocrine disorders (including diabetes, hypercholesterolemia, or dyslipidemia) that in the opinion of the Investigator would confound subject's participation and follow-up in the clinical trial.
2. Evidence of hepatorenal syndrome or acute glomerulonephritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentrations (Cmax) | from 0 hours to day 3
area under the plasma concentration versus time curve | from 0 hours to day 3

SECONDARY OUTCOMES:
Safety assessment with number of abnormalities reported by physical examination, vital signs,ECG, clinical laboratory parameters, local tolerability at injection site and adverse events. | Day 1-3 and day 1 of follow up visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami,Division of Clinical Pharmacology, Miami, Florida, United States

REFERENCES:
- [Derived] Preston RA, Mamikonyan G, DeGraff S, Chiou J, Kemper CJ, Xu A, Mastim M, Yeole R, Chavan R, Patel A, Friedland HD, Bhatia A. Single-Center Evaluation of the Pharmacokinetics of WCK 5222 (Cefepime-Zidebactam Combination) in Subjects with Renal Impairment. Antimicrob Agents Chemother. 2018 Dec 21;63(1):e01484-18. doi: 10.1128/AAC.01484-18. Print 2019 Jan. PMID 30397067